CLINICAL TRIAL: NCT06820541
Title: Prophylactic Endoscopic Transpapillary Gallbladder Drainage to Prevent Post-ERCP Cholecystitis After Covered Metal Stent Placement for Distal Biliary Obstruction: a Randomized Controlled Study
Brief Title: Gallbladder Stenting in FC-SEMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GB-COVER
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Biliary Obstruction; Acute Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be not informed about the treatment received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transpapillary stenting (Experimental): Patients will undergo prophylactic transpapillary gallbladder drainage followed by fully-covered self-expandable metal stent placement for biliary drainage
  Interventions: Device: Double plastic pigtail stent plus fully covered self-expandable metal stent
- Standard biliary drainage (Active Comparator): Patients will undergo fully-covered self-expandable metal stent placement for biliary drainage
  Interventions: Device: Fully covered self-expandable metal stent

INTERVENTIONS:
Device: Double plastic pigtail stent plus fully covered self-expandable metal stent — After contrast injection, the cystic duct orifice will be detected. Using a sphincterotome, a 0.035-inch hydrophilic angled guidewire will be negotiated into the gallbladder. Dilation of the cystic duct will be performed using standard devices designed for biliary intervention, including pneumatic dilators or dilation progressive catheters. After dilation, a 7Fr plastic, double pigtail stent, length of 12 or 15 cm, will be deployed across the papilla. Finally, a fully-covered self-expandable metal stent will be placed alongside the gallbladder drainage for biliary drainage.
  Arms: Transpapillary stenting
Device: Fully covered self-expandable metal stent — After biliary cannulation, a fully covered self-expandable metal stent will be placed for biliary drainage
  Arms: Standard biliary drainage

SUMMARY:
The goal of this randomized controlled trial is to determine whether primary prophylaxis with transpapillary gallbladder drainage prevents acute cholecystitis after fully-covered self-expandable metal stents placement during endoscopic retrograde cholangiopancreatography for malignant distal biliary obstruction in patients at higher risk of post-endoscopic retrograde cholangiopancreatography acute cholecystitis.

The main question it aims to answer is:

Does prophylactic transpapillary gallbladder drainage reduce the rate of post-endoscopic retrograde cholangiopancreatography acute cholecystitis in high-risk patients? Researchers will compare patients who undergo transpapillary gallbladder drainage to patients without transpapillary gallbladder drainage to see if transpapillary gallbladder drainage reduces the rate of acute cholecystitis.

Participants will:

1. receive or not transpapillary gallbladder drainage before fully-covered self-expandable metal stents placement
2. will be followed up at one, three, and six months to ascertain the onset of acute cholecystitis

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Signed informed consent
* Patients requiring covered metal stent placement for managing MBO
* High-risk of post-endoscopic cholangiopancreatography acute cholecystitis according to the following criteria:
* tumor involvement of the cystic duct orifice confirmed on magnetic resonance imaging, computed tomography, endoscopic ultrasound, or at endoscopic cholangiopancreatography;
* presence of at least 2 of the following:

  1. gallbladder stones;
  2. CBD diameter ≤ 10 mm;
  3. intraprocedural gallbladder opacification;
  4. cystic duct orifice at risk of being covered by the fully-covered stent

Exclusion Criteria:

* History of cholecystectomy
* Endoscopic retrograde cholangiopancreatography not feasible for duodenal stenosis or failed biliary cannulation
* Patients with previous gallbladder drainage
* Acute cholecystitis is already present based on the Tokyo guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Acute cholecystitis | 6 months
  The rate of acute cholecystitis, defined according to the Tokyo guideline, will be calculated and compared between the two groups

SECONDARY OUTCOMES:
Overall adverse events | 6 months
  The overall adverse events rate will be calculated and compared between the two groups
Hospitalization | 6 months
  The duration of the hospitalization will be calculated and
Disease-free survival | 6 months
  Acute cholecystitis free-survival rate, calculated as days from endoscopic retrograde cholangiopancreatography to acute cholecystitis or end of follow-up, cholecystectomy, or death, will be calculated and compared between the two groups
Technical success | 1 mont
  The rate of transpapillary gallbladder drainage, defined as the percentage of complete placement of the stent, will be calculated
Procedure time | 1 month
  The time of the procedure, calculates ad minutes starting after randomization to the end of the procedure, will be calculated and compared between the teo groups

CONTACTS AND LOCATIONS:
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No